CLINICAL TRIAL: NCT01991431
Title: Registry Of the Utilisation of the Transaortic (Tao) TAVI Approach Using the Edwards Sapien XT Valve
Brief Title: ROUTE Registry Of the Utilisation of the Transaortic (Tao) TAVI Approach Using the Edwards Sapien XT Valve
Acronym: ROUTE
Status: Completed | Type: Observational
Sponsor: Institut für Pharmakologie und Präventive Medizin (Network)
Responsible Party: Sponsor
Other Study IDs: U1111-1149-9900
Record Dates: First submitted 2013-11-06; First posted 2013-11-25 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TAVI: All Patients undergoing transaortic transcatheter valve implantation with commercially available Edwards SAPIEN XT Transcatheter Heart Valve with the Ascendra+ Delivery-System in participating sites

SUMMARY:
This is an international multi-center, prospective, observational registry with consecutive patient enrollment intended to determine outcome Parameters within 30 days after transaortic transcatheter aortic valve replacement.

DETAILED DESCRIPTION:
The purpose of this registry is to expand upon existing data sets, to identify patient characteristics and indicators related to complications and clinical benefits for patients with symptomatic severe calcific degenerative aortic stenosis that are undergoing transaortic transcatheter procedure with the commercially available Edwards SAPIEN XT Transcatheter Heart Valve with the Ascendra+ System.

ELIGIBILITY:
Inclusion Criteria:

* Intended transaortic (Tao) TAVI using Edwards SAPIEN XT Transcatheter Heart Valve with the Ascendra+ Delivery-System
* Compliance with the indications according to the Instructions for Use
* Written informed consent

Exclusion Criteria:

* Presence of contraindications as to the Instructions for Use
* TAo with concomitant procedure (e.g. Tao + CABG)
* Participation in the SOURCE XT registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Patients undergoing transaortic transcatheter valve implantation with commercially available Edwards SAPIEN XT Transcatheter Heart Valve with the Ascendra+ Delivery-System in participating sites
Sampling Method: Non-Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Overall mortality | 30 days
  to determine Overall mortality within 30 days after TAVI

SECONDARY OUTCOMES:
TAVI-related in-Hospital and 30 d mortality | 30 days after TAVI
  see title
complication rates | 30 days after TAVI
  Complication rates as to VARC2
Number of Patients with adverse Events in Relation to Baseline Parameters | 30 days after TAVI
  Identify multivariable adjusted predictors for adverse outcomes of transaortic TAVI

CONTACTS AND LOCATIONS:
Overall Officials: Vinayak Bapat, MD, Principal Investigator — St. Thomas' Hospital, London, UK; Mauro Romano, MD, Principal Investigator — Institut Hospitalier Jacques Cartier, Massy, France
Locations (19):
- Cardiac Surgery dpt., Innsbruck Medical University Hospital, Innsbruck, Austria
- Division of Cardiology, Helsinki University Central Hospital, Helsinki, Finland
- France (6):
  - CH J. Minjoz - Besancon, Besançon
  - CHU Bordeaux, Bordeaux
  - Hopital Cardio-Vasculaire et Pneumologie Louis Pradel, Lyon
  - Institut Jacques Cartier Massy, Massy
  - CHU Rouen, Rouen
  - CHU Rangueil - Toulouse, Toulouse
- Germany (4):
  - Robert-Bosch-Hospital Stuttgart, Stuttgart, Baden-Wurttemberg
  - Städt. Klinikum München GmbH Herzchirurgie Bogenhausen, München, Bavaria
  - Westdeutsches Herzzentrum Essen - Uniklinikum -, Essen, North Rhine-Westphalia
  - Universitätsklinikum Kiel - Kardiologie u. Angiologie, Kiel, Schleswig-Holstein
- Italy (2):
  - Univ. Padova, Azienda Ospedaliera di Padova, Padua
  - Policlinico San Matteo/Department of Cardiac Surgery, Pavia
- Academisch Medisch Centrum, Amsterdam, Netherlands
- Rikshospital Oslo, Oslo, Norway
- Klinika Kardiochirurgii UCK Gdansk, Gdansk, Poland
- United Kingdom (2):
  - St. Thomas Hospital Cardiothoracic surgery dept, London
  - James Cook Hospital - Cardiothoracic Division, Middlesbrough

REFERENCES:
- [Derived] Cocchieri R, Petzina R, Romano M, Jagielak D, Bonaros N, Aiello M, Lapeze J, Laine M, Chocron S, Muir D, Eichinger W, Thielmann M, Labrousse L, Rein KA, Verhoye JP, Gerosa G, Bapat V, Baumbach H, Sims H, Deutsch C, Bramlage P, Kurucova J, Thoenes M, Frank D. Outcomes after transaortic transcatheter aortic valve implantation: long-term findings from the European ROUTEdagger. Eur J Cardiothorac Surg. 2019 Apr 1;55(4):737-743. doi: 10.1093/ejcts/ezy333. PMID 30346515
- [Derived] Romano M, Frank D, Cocchieri R, Jagielak D, Bonaros N, Aiello M, Lapeze J, Laine M, Chocron S, Muir D, Eichinger W, Thielmann M, Labrousse L, Arne Rein K, Verhoye JP, Gerosa G, Baumbach H, Deutsch C, Bramlage P, Thoenes M, Bapat V. Transaortic transcatheter aortic valve implantation using SAPIEN XT or SAPIEN 3 valves in the ROUTE registry. Interact Cardiovasc Thorac Surg. 2017 Nov 1;25(5):757-764. doi: 10.1093/icvts/ivx159. PMID 28582580
- [Derived] Bonaros N, Petzina R, Cocchieri R, Jagielak D, Aiello M, Lapeze J, Laine M, Chocron S, Muir D, Eichinger W, Thielmann M, Labrousse L, Bapat V, Arne Rein K, Verhoye JP, Gerosa G, Baumbach H, Kofler M, Bramlage P, Deutsch C, Thoenes M, Frank D, Romano M. Transaortic transcatheter aortic valve implantation as a first-line choice or as a last resort? An analysis based on the ROUTE registry. Eur J Cardiothorac Surg. 2017 May 1;51(5):919-926. doi: 10.1093/ejcts/ezw406. PMID 28369303
- [Derived] Bapat V, Frank D, Cocchieri R, Jagielak D, Bonaros N, Aiello M, Lapeze J, Laine M, Chocron S, Muir D, Eichinger W, Thielmann M, Labrousse L, Rein KA, Verhoye JP, Gerosa G, Baumbach H, Bramlage P, Deutsch C, Thoenes M, Romano M. Transcatheter Aortic Valve Replacement Using Transaortic Access: Experience From the Multicenter, Multinational, Prospective ROUTE Registry. JACC Cardiovasc Interv. 2016 Sep 12;9(17):1815-22. doi: 10.1016/j.jcin.2016.06.031. PMID 27609256
- [Derived] Bramlage P, Romano M, Bonaros N, Cocchieri R, Jagielak D, Frank D, Bapat V. Transaortic transcatheter aortic valve implantation - rationale and design of the multicenter, multinational prospective ROUTE registry. BMC Cardiovasc Disord. 2014 Nov 1;14:152. doi: 10.1186/1471-2261-14-152. PMID 25361564
- See also: Design paper — http://bmccardiovascdisord.biomedcentral.com/articles/10.1186/1471-2261-14-152